CLINICAL TRIAL: NCT00683358
Title: Phase Ⅰ/Ⅱ Trial of Human Leukocyte Antigen (HLA)-A*2402-Restricted Vascular Endothelial Growth Factor Receptor 1 (VEGFR1)-Derived Peptide Vaccination Combined With Gemcitabine for Advanced Pancreatic Cancer
Brief Title: Human Leukocyte Antigen-A*2402-Restricted Tumor Vessel Specific Peptide Vaccination for Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tokyo University (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: Naohide Yamashita MD, PhD, Research Hospital, Institute of Medical Science, The University of Tokyo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMSUT-PPKVEGFR12402
Record Dates: First submitted 2008-05-16; First posted 2008-05-23 (Estimated); Last update posted 2009-05-07 (Estimated); Status verified 2009-01

CONDITIONS: Pancreatic Cancer; Pancreas Neoplasms
Keywords: cancer; pancreas; advanced; peptide; vaccination; VEGFR1; HLA; gemcitabine; IFA; Cancer of Pancreas; Neoplasms, Pancreatic; Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — HLA-A*24:02 antigen; Receptor Protein-Tyrosine Kinases; montanide ISA 51

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: VEGFR1-A24-1084 (SYGVLLWEI)

INTERVENTIONS:
Biological: VEGFR1-A24-1084 (SYGVLLWEI) — HLA-A*2402-restricted VEGFR1-derived peptide (VEGFR1-A24-1084) 1mg emulsified with Montanide ISA51 will be subcutaneously injected 2 times weekly for total 16doses concurrently with conventional dose of gemcitabine 1,000mg/m2 BSA on 1st, 2nd, 3rd, 5th, 6th, 7th weeks for advanced/inoperable pancreatic cancer patients.
  Other Names: HLA-A*2402; advanced pancreatic cancer; VEGFR1; VEGFR1-A24-1084; SYGVLLWEI; IFA; Montanide ISA51

SUMMARY:
Feasibility and efficacy of combined modality intervention using chemotherapeutic agent gemcitabine with anti-angiogenic peptide vaccination targeting VRGFR1 should be determined in case of advanced/inoperable or therapy-resistant pancreatic cancer patients.

Gemcitabine 1,000mg/m2 BSA will be administered on day1, day8, day15, day29, day36, day43, respectively.

HLA-A*2402-restricted VEGFR1-derived peptide (VEGFR1-A24-1084; SYGVLLWEI) emulsified with Montanide ISA51 will be subcutaneously injected twice weekly for 8weeks (total 16 doses).

DETAILED DESCRIPTION:
HLA-A*2402-restricted cytotoxic T lymphocyte (CTL) clones were obtained from healthy volunteer donor peripheral blood.

These CTL clones showed potent cytotoxicities selectively against VEGFR1-expressing target cells in HLA-class I-restricted manner.

ELIGIBILITY:
Inclusion Criteria:

* Heterozygote or homozygote of HLA-A*2402 allele
* Inoperable or recurrent pancreatic cancer with or without any prior therapy
* Difficult to continue the prior therapy due to treatment-related toxicities
* ECOG performance status 0-2
* Evaluable primary or metastatic lesion with RECIST criteria
* Clearance period from prior therapy more than 4 weeks
* Life expectancy more than 3 months
* Laboratory values as follows 2,000/μL<WBC<15,000/μL Platelet count>100,000/μL AST<150IU/L ALT<150IU/L Total bilirubin<3.0mg/dl Serum creatinine<3.0mg/dl

Exclusion Criteria:

* Pregnancy (refusal or inability to use effective contraceptives)
* Breastfeeding
* Active or uncontrolled infection
* Systemic use of corticosteroids or immunosuppressants
* Uncontrollable brain metastasis and/or meningeal infiltration
* Unhealed external wound
* Possibilities of complicated paralytic ileus or interstitial pneumonitis
* Decision of not eligible determined by principal investigator or attending doctor

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-04 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
PhaseⅠ; safety (NCI CTCAE v.3) PhaseⅡ；time to progression (RECIST) | 1 year

SECONDARY OUTCOMES:
Immune response (ELISPOT, Perforin/FoxP3 FACS, in vitro CTL assay etc.) | 1 year
Tumor regression(Imaging study, tumor marker, etc.) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Naohide Yamashita, MD, PhD, Study Director — Director, Research Hospital, Institute of Medical Science, Tokyo University
Locations (1):
- Research Hospital, The Institute of Medical Science, The University of Tokyo, Minato-ku, Tokyo, Japan

REFERENCES:
- [Background] Ishizaki H, Tsunoda T, Wada S, Yamauchi M, Shibuya M, Tahara H. Inhibition of tumor growth with antiangiogenic cancer vaccine using epitope peptides derived from human vascular endothelial growth factor receptor 1. Clin Cancer Res. 2006 Oct 1;12(19):5841-9. doi: 10.1158/1078-0432.CCR-06-0750. PMID 17020992
- [Background] Nagayama H, Sato K, Morishita M, Uchimaru K, Oyaizu N, Inazawa T, Yamasaki T, Enomoto M, Nakaoka T, Nakamura T, Maekawa T, Yamamoto A, Shimada S, Saida T, Kawakami Y, Asano S, Tani K, Takahashi TA, Yamashita N. Results of a phase I clinical study using autologous tumour lysate-pulsed monocyte-derived mature dendritic cell vaccinations for stage IV malignant melanoma patients combined with low dose interleukin-2. Melanoma Res. 2003 Oct;13(5):521-30. doi: 10.1097/00008390-200310000-00011. PMID 14512794
- See also: Related Info — http://www.transrec.jp/english/index.html